CLINICAL TRIAL: NCT04938544
Title: Determination of Insulin-stimulated Hepatic Glucose Uptake by PET-CT Measurements
Acronym: ISGU
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: NL74609.068.20
Record Dates: First submitted 2021-06-08; First posted 2021-06-24 (Actual); Last update posted 2023-03-29 (Actual); Status verified 2023-03

CONDITIONS: NAFLD; Insulin Resistance; Overweight and Obesity
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Insulin Resistance; Overweight; Obesity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — A fasting blood sample will be collected. Out of the fasted blood sample, DNA will be extracted from leucocytes in this sample to study genetic variants that may affect hormones and energy metabolism.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In the absence of excessive alcohol consumption, increased levels of fat in the liver (>5%) are diagnosed as non-alcoholic fatty liver (NAFL). It has been shown that NAFL is strongly associated with impairments in metabolic health such as hepatic and whole-body insulin resistance. Insulin resistance is seen as the earliest hallmark in the development of type 2 diabetes.

Insulin has two main effects on the liver: suppressing endogenous glucose production (EGP) and increasing glucose uptake. While the former has been extensively studied and is known to be impaired in NAFL, no studies have yet examined whether insulin-stimulated hepatic glucose uptake is affected by NAFL.

Recent methodological developments allow us to visualize and quantify glucose uptake in any given tissue using dynamic Positron Emission Tomography (PET) with 18Fluorinated glucose tracer (FDG) during insulin stimulation.

In the present study, we will in a first instance optimize the insulin-stimulated whole-body PET protocol and apply the dose as reported in the literature 4 megabequerels per kg of body weight (MBq/kg) (±8 mSv) in the first three subjects. It will then be evaluated whether the dose can be decreased in the remaining measurements. Another twelve individuals will then undergo the optimized dynamic PET protocol to assess insulin-stimulated hepatic glucose together with whole-body glucose uptake measures. Liver fat content and composition will be assessed by proton magnetic resonance spectroscopy (1H-MRS). Fasted De Novo Lipogenesis (DNL) will also be measured by deuterated water. Additionally, a two-step clamp will be performed to measure whole-body insulin sensitivity and insulin-stimulated suppression of EGP. The identification of the contributing factors to insulin resistance during the development of NAFL is crucial in order to develop more effective strategies for the prevention and treatment of metabolic disorders.

DETAILED DESCRIPTION:
Objective:

To determine the association between insulin-stimulated hepatic glucose uptake measured by dynamic PET and liver fat content in overweight/obese subjects.

ELIGIBILITY:
Inclusion Criteria:

* Caucasian (people will be excluded when having a ≥50% racial African/Asian background)
* Male or postmenopausal female
* Aged 45-75 years at start of the study
* Body mass index (BMI) 27 - 38 kg/m2
* Stable dietary habits (no weight loss or gain >3kg in the past 3 months)
* Sedentary lifestyle (not more than 2 hours of vigorous exercise per week)

Exclusion Criteria:

* Type 2 diabetes (fasted blood glucose > 7 mmol/L)
* Any condition or medical history that would in the investigator's or dependent physician's opinion interfere with the study, with study outcomes or increase the risk of the study procedures
* Alcohol consumption of >2 servings per day
* Smoking
* Low Hb (men: <8.6 mmol/L; women <7.4 mmol/L)
* Use of medication known to interfere with the safety of study procedures
* Use of medication known to increase liver fat, like for instance corticosteroids (parenteral & oral chronic administration only), amiodarone (Cordarone), tamoxifen (Nolvadex), and methotrexate (Rheumatrex, Trexall).
* Subjects receiving thiazolidinediones (glitazones [pioglitazone, rosiglitazone]).
* Participation in research or medical examination that included PET/CT scanning in the last 3 months
* Contra-indication for MRI

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A total of 15 healthy overweight/obese males and post-menopausal females (45-75 years, BMI 27-38 kg/m2) will participate in the study. Recruitment of participants will be performed in Maastricht and surroundings, by means of posters in public spaces (supermarkets, hospital, pharmacy, general practitioners), advertisements in local newspapers (e.g. Dagblad de Limburger and EenLokaal) and on the internet (e.g. digiprik.nl, proefbunny.nl and facebook.nl). Participants from previous studies will be contacted as well in case they provided written consent for this. To increase recruitment efficiency, potential participants can register at a mailing list. With this list, the researcher can approach individuals who showed interest in participating scientific research.
Sampling Method: Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2021-08-01 (Actual); Primary Completion 2023-05-31 (Estimated); Study Completion 2023-05-31 (Estimated)

PRIMARY OUTCOMES:
Insulin-stimulated glucose uptake measured by PET-CT measured by dynamic [18F]-FDG PET | 1 hour
  Insulin-stimulated hepatic glucose uptake rate constant (Ki) will be determined by [18F]- FDG PET, by using the Patlak method (Patlak et al. 1983) in each voxel. Influx rate will be calculated in mL/cm3/min
Hepatic fat content by 1H-MRS | 1 hour
  Liver fat will be quantified by 1H-MRS with which the water and fat resonances can be detected. The intensity of the fat resonance will be expressed relative to the water resonance (%).

OTHER OUTCOMES:
Hepatic insulin sensitivity measured by hyperinsulinemic-euglycemic clamp | 10 hours
  Hepatic insulin sensitivity is measured as % suppression of endogenous glucose production and peripheral insulin sensitivity is measured as Rd in μmol/kg/min. During the clamp, four blood samples in time are taken during each of the three steady states (basal, low insulin and high insulin phase). The average of these four blood samples will be taken for further calculations regarding glucose tracer kinetic: rate of appearance (Ra) and Rd.
Hepatic fatty acid composition by 1H-MRS | 1 hour
  Liver fat will be quantified by 1H-MRS with which the water and fat resonances can be detected. The intensity of the fat resonance will be expressed relative to the water resonance (%). Hepatic fatty acid composition is measured as relative amount of SFA, MUFA and PUFA to the total amount of fatty acids determined by MRS.
De Novo Lipogenesis | 1 day
  DNL is measured as relative contribution of newly synthesized palmitate in the VLDL-TG pool expressed as %DNL. The fasted blood sample will be used for determination of newly synthesized palmitate in the VLDL-TG pool.

CONTACTS AND LOCATIONS:
Overall Officials: Vera Schrauwen-Hinderling, PhD, Principal Investigator — v.schrauwen@maastrichtuniversity.nl
Locations (1):
- Maastricht University, Maastricht, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided